CLINICAL TRIAL: NCT04277286
Title: Non-randomized Experimental Study Evaluating the Impact of Implantation of a New Organization in the Adult Sector Intended to Improve the Transition of Young People With Endocrine or Metabolic Diseases
Brief Title: Evaluation of the TRANSEND Program
Acronym: EVATRANSEND
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP190984; IDRCB 2019-A02243-54 (Other: ANSM)
Record Dates: First submitted 2020-01-31; First posted 2020-02-20 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2021-02

CONDITIONS: Pediatric Patient Transfer to Adult Service:Transition Program
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental group: Patients transferred to adult service according to the Transend transition program (between September 2016 and January 2018)
  Interventions: Behavioral: survey
- Control group: Patients transferred to adult service without a transition program, in the same center, before the implementation of Transend (between January 2015 and September 2016)
  Interventions: Behavioral: survey

INTERVENTIONS:
Behavioral: survey — Behavioral study of patients who are in the "Transend" Program (compliance in follow-up visits after transfert from pediatric to adult care in the 24 months)

SUMMARY:
"Transend" is a program designed to promote the transition of young patients with endocrine or metabolic diseases when they arrive in the adult sector at La Pitié-Salpétrière hospital. The main objective of the study is to compare the rate of patients lost to follow-up at 24 months after the transfer of pediatrics between the Transend group and the (historical) control group.

DETAILED DESCRIPTION:
Adolescence and early adulthood represent important periods for young people suffering from chronic diseases. Several observational studies show needs not covered by care services at this period and significant lost to follow-up rates. "Transend" is a program designed to promote the transition of young patients with endocrine or metabolic diseases when they arrive in the adult sector at La Pitié-Salpétrière hospital (Paris, France). Since September 1, 2016, approximately 500 patients benefited from it.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 to 32
* Patient with endocrine or metabolic disease
* Patient who had a follow-up in a pediatric department for his endocrine or metabolic disease
* Patient transferred to the adult sector in the endocrinology, metabolism or nutrition department of Pitié-Salpêtrière
* Patient who had a first post-transfer consultation between January 1, 2015 and September 1, 2017
* Patient with a social security protection

Exclusion Criteria:

* Patient who transferred to another adult service before being followed at Pitié-Salpêtrière
* Patient who has expressed his opposition to participate in this research

Ages: 18 Years to 32 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Young patients with endocrine or metabolic diseases
Sampling Method: Probability Sample
Enrollment: 202 (Actual)
Dates: Start 2020-09-09 (Actual); Primary Completion 2020-10-10 (Actual); Study Completion 2020-10-10 (Actual)

PRIMARY OUTCOMES:
Rate of patients lost to follow-up at 24 months post transfert | 24 months post transfert
  Defined by pathology as patients who have not been seen in a medical consultation since a time superior of the recommendation for his state of Heath at 24 months post-transfer and for whom no elements confirm a next consultation in the center nor a follow-up in another center

SECONDARY OUTCOMES:
Number of consultations not honored by the patient | 24 to 36 months post transfert
  Experimental group: patients transferred to adult service according to the Transend transition program (between September 2016 and January 2018) Control group: patients transferred to adult service without a transition program, in the same center, before the implementation of Traansend (between January 2015 and September 2016)
Relationship of trust between caregiver and patient | 24 to 36 months post transfert
  Score calculated by wake Forest scaleis a validated scale of 10 items for the evaluation of the different components of trust.including 3 items on loyalty, 3 items on competence, 1 item on honesty and 3 items on global trust.
  (short version) resulting from an evaluation anonymously made by patients
Time to first consultation in adult medicine | 24 to 36 months post transfert
  Experimental group: patients transferred to adult service according to the Transend transition program (between September 2016 and January 2018) Control group: patients transferred to adult service without a transition program, in the same center, before the implementation of Traansend (between January 2015 and September 2016)
Patient satisfaction | 24 to 36 months post transfet
  Satisfaction collected on a scale of 0 to 10 where 0 means the worst transfer imaginable resulting an anonymous assessment carried out by the Patients
Avoided care consumption and associated costs | 24 to 36 months post transfret
  Costs associated with hospital emergency room visits, home visit of SOS doctor, unplanned hospitalization
Compare the experience of the transition betmeen the two Groups | 24 to 36 months post transfret
  Frequency of feeling broken, continuity, need to contact the paediatrician, attention and perceived availability on the part of professionals on arrival in the adult hospital
Assess Transend's efficiency | 24 to 36 months post transfret
  Cost/incremental cost-effectiveness ratio in cost gained and cost per loss of view

CONTACTS AND LOCATIONS:
Overall Officials: TOURAINE Philippe, PU-PH, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Chef du Service d'Endocrinologie et Médecine de le Reproduction, Hôpital de la Pitié-Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: No